

# **Using SMART Design to Improve Symptom Management Strategies Among Cancer Patients**

# National Cancer Institute Grant # 1 R01 CA193706 Study Protocol and Statistical Plan

May 28, 2020



# Research Strategy

# B. Significance

**1. Symptoms during Treatment: Solid Tumor Cancer Patients.** By 2030, cancer will surpass heart disease as the leading cause of death in the United States, with new cases expected to increase nearly 45% from 1.6 million to 2.3 million annually. Of highest significance to clinical practice, these patients are likely to experience the burden of symptoms resulting from cancer and its treatment, <sup>2-4</sup> leading to diminished health related quality of life (HRQOL). The adapted Barsevick symptom management model (Figure 2) guides this study. Based on the model, improved symptom management, especially fatigue, is the proposed mechanism for improving HRQOL.

Symptoms are defined as patient's perceptions of abnormal emotional and physical states. 11

<u>Primary Outcome</u>: Fatigue is the most prevalent and often distressing symptom related to cancer and its treatment. <sup>12</sup> The prevalence of cancer-related fatigue during active treatment



ranges from 25% to 99% based on the sample and methods of assessment. 13 Cancer-related fatigue is the perception of unusual tiredness that varies in pattern and severity and has a negative impact on ability to function in people who have or have had cancer. 10 Due to the high prevalence of fatigue

and this team's completed work showing efficacy of two interventions for this symptom,<sup>5,14</sup> fatigue is the primary outcome of the proposed study. Fatigue is known to affect HRQOL outcomes.<sup>10,15-20</sup> The biological changes due to chemotherapy and the resulting inflammatory processes may be responsible for the persistence of fatigue, as well as related symptoms.<sup>21-23</sup> Physical, emotional and cognitive components of fatigue will be captured in this study.

Secondary Symptom Outcomes: In a survey of a 1000 cancer patients, the mean number of symptoms reported was eleven.<sup>24</sup> Therefore we will evaluate three secondary outcomes: 1) summed severity score across an array of symptoms other than fatigue (to avoid duplication with primary outcome) from the expanded M.D. Anderson Symptom Inventory (MDASI)<sup>25,26</sup> pain, nausea, disturbed sleep, distress, shortness of breath (dyspnea), difficulty remembering, decreased appetite, drowsiness, dry mouth, sadness, vomiting, numbness/tingling, cough, constipation, diarrhea, sore mouth, rash, and hair loss; 2) depressive symptoms; and 3) anxiety. A key symptom example from the MDASI is dyspnea, a multidimensional subjective experience of breathing distress that impairs functional status, and is associated with thoughts about

disability, lowered hopefulness, and existential problems in individuals with cancer.<sup>27,28</sup> In our completed studies with reflexology and meditative practices, there was a significant improvement in self-reported dyspnea.<sup>5,29</sup> We will also assess two symptoms not specifically included in MDASI: depression and anxiety that are common in cancer patients and are a source of high distress and decrease in HRQOL.<sup>30,31</sup> Our preliminary data,<sup>32,33</sup> published work,<sup>5,14</sup> and work of others<sup>13,26-30</sup> indicate the interventions we propose in this study may impact primarily fatigue, but also dyspnea, depression and anxiety.<sup>14,26,34-37</sup> One primary and three secondary outcomes evaluated in this study will reflect the burden of multiple symptoms that cancer patients experience.

2. Home-Based Symptom Management with Caregivers. This project is also significant because it meaningfully engages a friend or family member in their patients' supportive care over time. Many randomized controlled trials (RCT) of symptom management interventions. including complementary therapies, consist of an intervention period of several weeks, which does not cover the full duration of cancer treatment. Since symptom management is needed not just for a few weeks, but for the entire cancer treatment and beyond, the engagement of a friend or family caregiver may represent a significant solution to the sustainability of home-based symptom management interventions. In our nearly completed R01 with reflexology for cancer symptom management, we engage friend or family caregivers.<sup>33</sup> A friend or family caregiver is identified as such by the patient and provides unpaid assistance to a person with a chronic or disabling condition such as cancer.<sup>38,39</sup> Currently, the estimated number of cancer patient caregivers is 5.7 million people. The value of this unpaid labor force of caregivers in the U.S. 40,41 is appraised to be at least \$306 billion annually. 42,43 It is recognized that the support provided by caregivers may influence the outcomes of their patient's cancer treatment. 38,44-46 Caregivers may also be an important influence on patient care options since they are key stakeholders in patients' symptom management. In this sense, interventions that support the patient may also indirectly support the caregiver. 47,48 For these reasons, our project targets the caregiver along with the patient to engage in the home-based symptom management intervention/s.

Home-based Interventions. Despite the high needs for symptom care, patients undergoing cancer treatment have limited choices, given their unique vulnerabilities.<sup>49</sup> Reduced functional status can lead to difficulties with the use of supportive therapies that require travel or a group format.14 Further, patients with symptoms such as dyspnea are at a higher risk due to weather changes, another factor which reduces function and accessibility to interventions that are provided outside the home.<sup>27,37</sup> While home-based interventions during cancer treatment are potentially significant, many do not produce clinically or practically meaningful improvements. For example, while the effects of supervised exercise interventions on the improvement in fatigue are moderate to large (e.g., d=0.75-0.87<sup>50</sup> and d=0.95-1.00), <sup>50-52</sup> the effects of homebased unsupervised exercise interventions are generally small,<sup>53</sup> with standardized mean difference for high-quality studies in meta-analysis being as small as 0.13.52 Further, limited evidence from quality randomized trials exists to support the use of dietary supplements for fatigue during chemotherapy, with dietary counseling being more promising compared to supplementation. When bundled with exercise interventions, the added benefit of dietary advice does not appear to increase the effect sizes, compared to those reported from exercise interventions alone.<sup>54</sup> Supervised exercise interventions bundled with dietary advice produce moderate to large effect sizes, 55 and self-directed home-based bundled interventions produce small effect sizes. 56-58

Home-based symptom management interventions in this study, reflexology and meditative practices, have been tested against controls and attention controls in randomized controlled trials, and have been shown to produce moderate to large effect sizes (see preliminary work).<sup>5,32</sup> Each home-based intervention provides a significant strategy to manage fatigue during chemotherapy. However in practice, individual patients vary in their responses to interventions and may try various combinations of symptom management strategies.<sup>59</sup> So the next innovative step after establishing efficacy against controls is individualization and sequencing of interventions using the SMART design.<sup>60,61</sup> The two interventions considered in the proposed research use different approaches; one is physical (reflexology) and one psychological (meditative practices). Therefore the success of these interventions may be different for different patients, and there is a need to either lengthen the time with one therapy or test the effects of adding a different therapy when one does not produce the desired outcomes in a given period of time. The SMART design provides a rigorous framework for such testing because of the strength of conclusions that will be derived from randomized comparisons.

3. Interventions: Two Complementary and Alternative Medicine (CAM) Therapies. An increasing number of cancer patients turn to CAM therapies for symptom management.<sup>62</sup> Our team's program of research focuses on building the evidence base for CAM that may enhance symptom management among cancer patients, in order to determine which therapies warrant translation to practice, and which elicit comfort or placebo effects but do not add to the pool of effective symptom management interventions.<sup>63</sup> The widespread use of complementary therapies in patients is exemplified by a significant increase (p≤.001) over a 7-year time span for common chronic conditions. 64 The National Health Interview Survey reported that 38% of Americans use some type of complementary therapy. 65 The highest users of CAM therapies are younger adult females. 66 Additional factors associated with CAM use vary across studies and include higher education, private insurance, regular exercise, or attending support groups. 66-70 Surveys have found that over time more minority patients are using CAM, with some variation on the types of therapies selected by racial and ethnic underrepresented. 67,68,71 Recent literature also indicates high prevalence of CAM use among men and in low-income urban minority populations. 66 When complementary therapies are used by the public to this extent and without adequate knowledge of safety and efficacy, they run the risk of interfering with conventional health care. Therefore, before complementary therapies can become part of evidence-based symptom management practice, they need to be rigorously tested in RCTs against controls and other therapies, and evidence-based decision rules for best selections and sequences of therapies need to be determined.

The National Center for Complementary and Alternative Medicine (NCCAM)<sup>72</sup> identified five categories of complementary therapies: mind-body; body-based; biologically based; energy therapies; and alternative medical systems. **We have selected a body-based therapy and a mind-body therapy because these two therapy groups are the most widely used by cancer patients,**<sup>73</sup> provide different approaches, and both have a demonstrated evidence base against controls.<sup>5,14,74,75</sup> This evidence is summarized below.

<u>Reflexology</u>. Reflexology is similar to massage in that it manipulates soft tissue for therapeutic purposes, but differs due to the focus on the special areas of the feet called reflexes and the use of a firm thumb-walking motion.<sup>76</sup> It is based on the premise that foot reflexes correspond to organs, glands, and body systems. Stimulating these reflexes may positively affect function of

the target tissue to facilitate health and healing. 76 Current research regarding the impact of reflexology on symptom management is burgeoning.<sup>5</sup> Our team's completed R01 (5R01CA104883-5) demonstrated a significant decrease in fatigue when foot therapy was provided by a lay caregiver.<sup>5</sup> A systematic review of RCTs<sup>77</sup> found that in two cancer studies, reflexology resulted in a significant decrease in anxiety.<sup>78</sup> and a significant improvement in QOL.<sup>79</sup> A second review<sup>80</sup> demonstrated an immediate post-intervention reduction in pain. Since these systematic reviews, five RCTs focused on a cancer patient population. One study reported significantly lower anxiety among multiple types of cancer patients, 81 another found lower pain with a mixed cancer group. 82 a third reported decreased pain among digestive cancer patients, 83 a fourth, using a bundled intervention, found that eight weekly sessions of reflexology plus self-initiated support significantly promoted relaxation among post-surgical early-stage breast cancer patients (n=60).84 and a fifth study involved a mixed sample of hospitalized cancer patients (n=42) where a partner provided one session, resulting in an immediate decrease in pain intensity and anxiety.<sup>74</sup> Our team completed the first large scale RCT with reflexology (n=385 breast cancer patients), and demonstrated a significant improvement in physical functioning and dyspnea following 4 weekly sessions by a reflexologist. The results from the completed RCT of reflexology and the preliminary results from our nearly completed trial (1R01CA157459-01), where reflexology is delivered by a friend or family caregiver, are presented under justification and feasibility.

Reflexology is a significant body-based intervention selection because it: 1) is non-invasive; 2) extremely low risk; 3) does not interfere with cancer treatment the patient is receiving;<sup>5</sup> 4) can easily be taught in the home to a friend or family caregiver;<sup>33</sup> and 5) based on a national survey, patients are highly likely to use it.<sup>85</sup>

<u>Meditative Practices.</u> Meditative practices are purposeful strategies aimed towards building capacities to attend to the present moment, including one's thoughts, emotions, bodily sensations, and the environment with nonjudgmental openness and acceptance.<sup>86</sup> This therapy selection is grounded in evidence that meditation training with gentle yoga and breathing exercises enhance patients' ability to adapt to serious medical concerns.<sup>87-91</sup>

In our completed work presented under justification and feasibility, teaching meditative practices demonstrated feasibility, acceptability and efficacy for symptom management among lung cancer patients. 14,32 Studies that incorporate meditation-based therapies in cancer are increasing and are showing promise in modifying psychological distress and improving HRQOL. 92-94 Such research in cancer groups include studies incorporating observational, 35,95-97 non-randomized prospective experimental, 98,99 and RCT designs. 100-104 Studies in cancer report that training in meditative practices resulted in significant improvements in mood, 105,106 anxiety 31,75,97,101,105,107, depression, 31,75,101,108 fatigue, 36,102,105 HRQOL, 75,98,101 stress, 97,101,108,109 coping, 97,109,110 and sleep quality. 96,99,104 In two RCTs, engagement in meditative practices reduced perceived stress, 103 and psychological distress, 75,105 demonstrating efficacy in modulating emotional symptoms.

Meditative practices are a significant mind-body intervention selection because they: **1)** have been tested with solid tumor cancer patients; <sup>97-99,101,104,110</sup> **2)** are a highly-utilized supportive therapy with vulnerable cancer patients; <sup>75,93</sup> **3)** have been shown to promote adjustment, reduce psychological distress, and improve HRQOL in cancer patients; <sup>94,109</sup> **4)** are economically delivered and feasible for patients to use on their own at home; <sup>94</sup> and **5)** are a non-toxic option for symptom management during active treatment.

Rationale for sequencing of therapies (reflexology and meditative practices). While there are likely several physiological mechanisms involved that contribute to the positive outcomes from reflexology and meditative practices, the benefits derived from reflexology, a direct body manipulation are primarily physically mediated; whereas, the effects derived from training in meditative practices are cognitively-mediated. 91 Reflexology has been implicated in the activation of oxytocin, and to optimize circulatory capacity to eliminate toxins and support immune, nervous, and glandular systems. 84,111 In Magnetic Resonance Image brain scans, meditative practices have demonstrated growth in brain regions that are involved in emotion regulation, attention, learning, and memory function. 112 Both reflexology and meditative practices result in activation of a relaxation response<sup>84,111</sup> characterized by calmness, sensations of wellbeing, and acceptance which may contribute to heightened HRQOL. We will test one therapy, and if it is inadequate, we will either: 1) add the alternative therapy -recognizing that an alternate therapy may evoke benefits by targeting another pathway to yield the sought benefits, or 2) provide a longer duration of the first therapy. Because of these potential systemic effects, the benefits of reflexology and meditative practices are not limited to immediate results and may be cumulative over time. Therefore extending duration of a single therapy is one possibility to achieve desired symptom reduction. On the other hand, the use of two therapies, that evoke the relaxation response via different pathways to gain similar symptom management, may optimize the potential for therapeutic benefits. Some people may prefer or respond better to a cognitive therapy over direct physical contact, while others may favor bodybased reflexology, and the optimal intervention choice and sequencing may depend on such individual differences. The SMART design allows for rigorously testing and tailoring intervention sequences to patients.

4. SMART Design. Existing static symptom management interventions deliver a predetermined dose at specific intervals. These interventions are tested in standard RCTs against controls, and this has already been done for reflexology and meditative practices. Dynamic tailoring of interventions to patient responses is needed to enhance the science of symptom management. 113,114 This gap in science is filled by the SMART design in which we will test interventions that target symptom severity and adjust intensity based on patient response to the management of fatigue. Our approach builds sequences which start with one therapy, and then at a decision point, symptom response is evaluated and one intervention may continue so as to give it more time, or the intervention is intensified by adding a second therapy. If one therapy of 4 or 8 weeks is successful, this information is important for both patient and caregiver who can then target the one best therapy. Other dyads may need the intensity of two therapies. In this case, an important question is whether it is best to start with reflexology or with meditative practices and then add the second therapy, and the proposed research will assess which patient and caregiver characteristics are important in making this decision for future work. While SMART designs do not typically include a control group (since first and second stage interventions have been pre-tested in standard RCTs), we included one to help gauge the clinical significance of improvements in symptoms from sequences of interventions that originate from the first randomization. The evidence obtained in the analysis of the intervention sequences will guide refined algorithms for allocating intervention resources in a way that leads to the best possible patient outcomes.



#### C. Innovation

The key innovations that maximize the potential of the intervention sequences to improve symptom outcomes are:

- 1. Involvement of a friend or family caregiver in delivery of a multistage home-based intervention for symptom management over time. Family involvement has been a missing link in sustaining home-based symptom management. Many interventions require delivery by a provider outside of the home and can be expensive. This research creatively utilizes a multistage intervention that builds on evidence established in our work that friend or family caregivers can successfully learn to deliver reflexology and can also participate and/or support patients with their meditative practices over time in nonclinical environments such as the patient's home.
- **2. Rigorous investigation of combinations and sequencing of therapies.** Past research on complementary interventions often bundled several therapies together, and the resulting outcomes could not be attributed to specific therapies. The proposed study takes a new approach to the rigorous testing of the value added by a second therapy if the first one does not achieve outcomes. The step-up approach with the second randomization provides a design where the effect of intensifying an intervention with a second therapy versus giving a single therapy more time (higher dose) can be isolated.
- 3. Dynamic delivery model and cutting-edge statistical methods. The innovative SMART design allows us to investigate the sequencing of interventions based on their success with individual patients. Designs similar to SMART have begun to be implemented in chronic conditions 119-122 including cancer, 123,124 and their use for optimizing behavioral interventions has been suggested in PA-13-165<sup>125</sup>that we are responding to. **To our knowledge, this research** is the first to use the SMART design for symptom management in cancer patients. This innovative dynamic delivery model is ideally suited for the temporal nature of symptoms that present challenges to symptom management science. 11,126-128 The exploratory Aim 5 analyses use a Q-learning algorithm to determine optimal decision rules for choosing intervention sequences for individual patients in the future, based on their characteristics and the characteristics of the caregivers who will be providing these home-based interventions or practicing them with the patients. The Q-learning algorithm allows for inclusion of time-varying covariates, 129 such as repeated measures of symptom severity at baseline and over the first 4 weeks, to determine if adding another intervention during weeks 5-8 is warranted. The resulting new clinical decision rules and algorithms have the potential to optimize the delivery of supportive care interventions given individual dyadic profiles.

# D. Approach

# 1. Justification and feasibility

<u>1a. Preliminary Work with Patient Selection of Therapy.</u> In preliminary work, our team administered a 25-item complementary therapy survey to 27 cancer survivors. Strong interest was shown for both mind-body therapies such as meditative practices and body-based physical touch therapies such as reflexology.<sup>130</sup>

We then conducted a quasi-experimental study with 100 mixed cancer patients in active treatment to participate over eight weeks with a family caregiver. Results demonstrated acceptability and feasibility of caregiver participation in complementary supportive therapies.<sup>131</sup>

1b. Preliminary Work with Reflexology. In our recently completed reflexology RCT with 385 women in treatment for breast cancer, no adverse events were reported, and > 89% of women in the reflexology group completed three or four sessions of the four session protocol. Longitudinal comparisons revealed significant improvements in physical functioning for the reflexology group compared to the control group (p=.04). Dyspnea severity was reduced compared with the control (p < .01) and lay foot manipulation (LFM) groups (p = .02). The effects sizes for the improvements in dyspnea and physical function in the reflexology group compared to controls and LFM were medium to large (between 0.41 and 0.87 for average differences between groups over time). No differences were found for depressive symptoms or state anxiety. The LFM group had a significant improvement in fatigue compared to controls (p=.01).

1c. Preliminary Work with Reflexology and Caregivers. In the principal investigators' (PIs) ongoing R01, both patients and their friend or family caregivers are enrolled as dyads in a reflexology study for symptom support and reduction of unscheduled health services used. We have been successful in maintaining scheduled dyad enrollment (N=240 consented and 190 randomized after completing baseline interview as of February, 2015). Friend and family caregivers have been able to achieve protocol proficiency at 90% immediately after training and at the follow-up quality assurance check a week later. 132

| Table 1. Preliminary Work: Reflexology and Caregivers | | | | |
|---|---|---|---|---|
| | Caregiver-<br>delivered<br>reflexology<br>LS Mean (SE)<br>N=72 | Attention<br>control<br>LS Mean<br>(SE) N=68 | P-<br>value | Effect<br>size |
| Fatigue severity | 3.64 (0.23) | 4.32 (0.23) | .04 | .46 |
| Insomnia severity | 2.95 (0.26) | 3.57 (0.27) | .10 | .31 |
| Pain severity | 2.25 (0.23) | 3.21 (0.24) | <.01 | .49 |
| MDASI total symptom severity | 25.07 (1.59) | 30.63 (1.63) | .02 | .48 |
| MDASI total symptom interference | 12.15 (1.15) | 16.08 (1.17) | .02 | .48 |

After caregiver training, the rate of protocol completion is high for more than one session per week (69%, 89%, 82%, and 83% by week). Virtually all dyads that completed at least one session actually did 2 or more, which indicates the willingness and interest of caregivers in delivering reflexology sessions

to patients. Outcomes are measured at baseline, week 5 (post 4-week intervention) and at 11 week follow-up. Analysis included group comparisons at weeks 5 and 11 using linear mixed effects models and estimation of the effect sizes (Cohen's d) for average group differences over time expressed in standard deviation units. The results from N=140 dyads who completed the 5 and/or 11 week interview to date are summarized in Table 1. P-values <.05 and clinically significant effects sizes >0.33 are bolded. The significant improvements due to caregiver-delivered reflexology are seen in severity of fatigue, pain, and summed symptom severity and interference (MDASI).

<u>1d. Preliminary work with meditative practices.</u> To develop our meditative practices intervention, we first conducted focus groups with cancer patients who had undergone radiation (RT) and chemotherapy.<sup>14</sup>

Table 2. Preliminary work with Meditative Practices

| | Meditative<br>practices<br>LS Mean (SE) | Attention<br>control<br>LS Mean (SE) | P-<br>value | Effect<br>size |
|---|---|---|---|---|
| SF-36 Vitality (lack of fatigue) | 47.92 (2.19) | 44.15 (2.06) | 0.24 | 0.45 |
| Total Dyspnea Score | 3.64 (1.07) | 7.60 (0.99) | 0.02 | 0.96 |
| SF-36 Bodily Pain | 48.89 (2.39) | 44.93 (2.25) | 0.26 | 0.41 |
| Cancer Worry | 6.17 (0.53) | 8.07 (0.49) | 0.02 | 0.85 |
| Depressive symptoms (CESD) | 7.84 (1.80) | 12.76 (1.68) | 0.07 | 0.70 |
| Sleep Quality Problems | 8.38 (1.87) | 11.76 (1.75) | 0.22 | 0.45 |

Based on the findings from these focus groups, we developed a shortened home-based intervention responsive to the needs of vulnerable cancer patients who are in treatment. The adapted meditative practices protocol was tested with 40 patients with lung cancer [mean age:

66.2±9.4 years; sex: 27(67.5%) females, 13(32.5%) males; disease stage: III, 10(25%); IV, 30(75%)] receiving radiation and/or chemotherapy. Patients were randomized to receive weekly meditative practice sessions (N=20) or an attention control condition (N=20). Outcomes were measured at baseline, post intervention and at 11 weeks. Table 2 summarizes the least squares (LS) means, their standard errors (SE), p-values and adjusted effect sizes for group comparisons. Due to relatively small sample size, statistical significance was not reached for all outcomes; however the effect sizes indicate clinically significant improvements and the magnitude of the effect sizes is similar to those seen in Table 1 for the reflexology intervention. The study demonstrated feasibility of our adapted meditative practices program, and early efficacy with respect to symptom reduction. <sup>32</sup>

2. Team. Our team is led by Co-PIs Drs. Gwen Wyatt and Alla Sikorskii. Dr. Wyatt is a professor in the College of Nursing, whose research program focuses on testing complementary therapies as supportive care interventions for cancer patients to lessen symptoms and enhance HRQOL. 130,131,133-142 She is currently PI on a NCI 1R01 (CA 157459-01) involving reflexology and a friend or family caregiver; she is also Co-I on an acupressure study with breast cancer survivors (1R01 CA151445-03); and has completed a reflexology RCT (1R01 CA104883-01A1) with breast cancer patients. Dr. Sikorskii is an associate professor in the Department of Statistics and Probability, statistician and methodologist who has collaborated with Dr. Wyatt since 2004 and is currently a Co-Investigator (Co-I) on the ongoing reflexology R01. In addition to the ongoing reflexology RCT, Dr. Sikorskii has served as a Co-I on 10 NIH funded R01 grants and one large CDC-funded study. The multiple PI leadership is essential to the proposed project that requires expertise in symptom management and complementary interventions as well as expertise in design and methodology of intervention testing. Co-I Dr. Rebecca Lehto is an assistant professor and expert oncology clinician who investigates meditative practices in cancer patients to facilitate improvement of cognitively-mediated symptoms. Our team consultants are: Elizabeth Marazita, a Doctor of Oriental Medicine and reflexology expert; and Denise Kozikowski, PhD who is a psychologist and certified expert in meditative practices.

Other Personnel. Recruiters will be located at each site. Interviewers will contact participants via telephone at baseline and week 12 from the main research office. Intervention experts will train and QA the study reflexologists and meditative practices teachers; study reflexologists will train caregivers in reflexology and meditative practices teachers will train caregivers in meditative practices. The Education Coordinator (EC) will schedule and coordinate all training, and make weekly calls to caregivers.

**3. Setting.** We will begin with 3-4 oncology clinics in the Midwest, and open additional sites if needed to maintain enrollment. All dyad therapy sessions will be done in the home.

**4. Sample.** Patients will be approached at the participating oncology clinics. Inclusion criteria are: 1) age 21 or older; 2) solid tumor cancer diagnosis; 3) able to perform basic activities of daily living; 4) undergoing chemotherapy, hormonal therapy, or targeted therapy; 5) reporting severity of ≥3 on fatigue using a 0-10 standardized scale at intake; 6) able to speak and understand English; 7) have telephone access; and 8) able to hear normal conversation. Exclusion criteria are: 1) diagnosis of major mental illness in medical record and verified by the recruiter; 2) nursing home resident; 3) bedridden; 4) currently involved with reflexology or meditative practices; or 5) deep vein thrombosis or painful foot neuropathy.

Solid tumors have been selected because fatigue can be effectively managed with the two interventions based on existing evidence, and this symptom is prevalent during cancer treatment. The cut-off of  $\geq 3$  indicates a moderate level of fatigue based on established interference-based cut-points. Virtually all solid tumor cancer patients on chemotherapy reach a threshold of 2 or higher on fatigue at some point, and the cut-off of 3 was found to be optimal in past work for balancing sensitivity and specificity in the prediction of the need for symptom management in the future 8 weeks. Weeks.

Friends/family caregivers will participate with each patient and will complete a consent form. Their inclusion criteria are: 1) age 18 or older; 2) able to speak and understand English; 3) access to a telephone; 4) able to hear normal conversation; 5) cognitively oriented to time, place and person (determined via recruiter); and 6) willing to be trained in reflexology and meditative practices.

- 4a. Sample size. To determine the sample size for this study, we started at the right end of the schematic in Figure 1 (the second randomization) and moved from right to left to determine the needed number of consenting patients. To power the comparisons for the value added by reflexology or meditative practices, we used the effect size of 0.45, the smaller of the two effects sizes for fatigue from Tables 1 and 2 to conservatively estimate sample size requirements. The effect size of 0.45 corresponded to 2 repeated measures in past work, and the design of this study includes 4 repeated measures at each phase. Assuming a correlation of 0.4 among repeated measures seen in past work, the adjusted effect size for the longitudinal analysis of 4 time points is 0.54, which results in the sample size requirement of N=55 per group being compared (far right of Figure 1), for power of .80 or greater in two-tailed tests at 0.05 level of significance. These 55 patients from 4 groups (220 total) created by the second randomization will be non-responders from the first intervention stage. Assuming that these 220 are 80% of the total number of patients in the first stage (i.e., that there is a 20% response rate to fatigue during the first 4 weeks), we will need 276 patients to be randomized to interventions. The size of the control group was selected to be 55 to maximize power in the comparisons with intervention subgroups. Therefore the total required post-attrition sample size is N=331. To account for 23% attrition seen in past work<sup>5,147</sup> with solid tumor cancer patients, we will need to have 430 patients consent.
- 4b. Strategies to minimize sample attrition. 1) Recruiters will emphasize the importance of participating in the full intervention and the weekly calls; 2) patients will be asked to mark their home calendar for intervention days and study calls; and 3) weekly calls to patients maintain contact for the entire study duration. These strategies have worked well in our completed and ongoing trials.

- Participants will be assured of the confidentiality of all information and that refusing to participate will not alter their care. Patients will continue to receive standard medical care, so if any healthcare problems arise, they may seek care from their health providers. For patients who refuse, the recruiter will seek consent to review their record for demographics and ask the reason for refusal. These data help us understand who declines and contribute to external validity and generalizability of the findings.
- **5. Recruitment.** Our team has an existing relationship with 14 oncology clinics in the Midwest. Even with recruitment challenges, <sup>148</sup> we are confident of achieving the recruitment target of 430 before attrition, and a post-attrition sample size of 331. In our recently completed reflexology R01 (N=385 breast cancer patients), we were able to remain within 10% of recruitment goals for the four years of enrollment and had a consent rate of 74%. In our current R01 with both cancer patients and their caregivers (planned N=200 patients; 200 caregivers post-attrition), we are having similar enrollment rates during year four. As of February 2015, N=190 dyads have completed baseline interview and were randomized. Our samples are representative of the cancer patient populations in the Midwest. In the most recent reflexology trial, 14% of patients and 13% of caregivers were African American, and 4% were Hispanic. <sup>33</sup>
- <u>5a. Accrual.</u> Recruiters have research roles and do not provide direct care at the sites. They will approach patients during clinic visits and explain the study. Patients can choose to consent at that time if their caregiver is present, or take the packet home to discuss with their caregiver. Recruiters will follow up during a clinic visit or by phone to further explain the study, answer questions, and discuss the study with caregivers. If verbal consent is obtained over the phone for either the patient or caregiver, the consent forms in the packet can be signed and returned in the stamped envelope. If the consent forms are not returned within one week, the recruiter will call as a reminder to mail the consent forms if they wish to participate.
- <u>5b. Recruiter training</u> includes didactic information, role-playing, problem cases and return-demonstration conducted by the study Education Coordinator at sites. Recruiters will use a script to introduce the study to patients including: 1) initial randomization to reflexology, meditative practices for symptom management or a usual care control group, and the possibility of the two active groups being re-randomized after 4 weeks of using the first therapy to either continue the same therapy or to also add the other therapy; 2) weekly intervention sessions provided by their caregiver in the two active groups (following training by a reflexologist and/or a meditative practices teacher) in their home; 3) there is no cost; 4) the complete study lasts 12 weeks to include all data collection (i.e., weekly calls and two 30-45 minute phone interviews); 5) both therapies are designed to help reduce symptoms and improve HRQOL; and 6) a review of potential risks/benefits.
- **6. Randomization.** Following the baseline interview, patients will be randomized to reflexology, meditative practices or standard care control. Randomization will be completed using a computer minimization algorithm programmed by Dr. Sikorskii that balances arms by recruitment location, site of cancer, stage of cancer (early versus late) type of treatment (chemotherapy, hormonal therapy or targeted therapy, and their combinations), patient sex and relationship to the caregiver (spouse vs non-spouse). The second randomization will occur for those who do not respond on fatigue to the therapy received after the first 4 weeks of therapy. The second randomization will be implemented using the same approach as the first, with the same balancing factors, except that randomization will allocate patients into 2 groups: continuing the same therapy or adding the other one.



# 7. Intervention Components

<u>7a. Active Group Caregiver Intervention Procedures.</u> Caregivers will: **1)** be trained by a study reflexologist or meditation teacher in the therapy their patient is initially randomized to; **2)** after 4 weeks of delivering the therapy, caregivers will be trained in the second therapy if their patient is re-randomized to receive the other therapy; **3)** receive weekly calls over 8 weeks to maintain fidelity and inquire about the number of sessions completed in the past 7 days. At least one weekly session is required per protocol. The number of additional sessions per week is not restricted in a home-based intervention, and the number of sessions delivered is tracked weekly (see 7d, Protocol Fidelity).

<u>7b. Intervention Protocols.</u> As recommended by the NCCAM, complementary therapy investigators should partner with therapy experts, while acknowledging that the investigator role requires very different preparation than that of the practitioner. Our team has successfully maintained this role delineation and will again engage leading experts to assure protocol fidelity and delivery. Consultant Dr. Elizabeth Marazita, reflexology expert, will oversee the protocol via start up and annual consultation with Dr. Wyatt and our training reflexologists. Consultant Dr. Denise Kozikowski, meditative practices expert, will oversee the protocol via start up and annual consultation with Co-I Dr. Lehto and our training meditation teacher (see experts & trainers letters of support). The consultants and trainer for each therapy will have no direct contact with participants; this further assures protection against contamination of roles.

7c. Common Elements to Study Provider Training. The intervention trainers will train the study providers who will work directly with patients and caregivers. Study provider reflexologists will be practicing reflexologists, who will be trained in the study specific protocol. Study meditation providers will be health professionals, e.g., nurses. Training for both therapies will include didactic information, written steps of the protocol, role-playing, demonstrations, and return-demonstrations based on our study-specific criteria. All study providers must demonstration protocol proficiency ≥ 90% to begin and continue (QA checks) with participants (proficiency check list in appendix). Both therapies have written instructions with diagrams that will be left with caregivers. In addition, to enhance the utilization of technology, a DVD demonstrating the instructions will be offered to all dyads. Each study provider will be in the home approximately 45-60 minutes during the first two weeks of the caregiver using the therapy. The first visit is for training and the second to observe and smooth out any errors. This method of caregiver involvement is working well in our ongoing R01.<sup>132</sup> All caregivers will be expected to involve the patient in a minimum of one session per week. Study providers will help the patient and caregiver select a day and time each week for the home-based session.

7d. Protocol Fidelity and Number of Sessions Per Week. Intervention protocol fidelity will be assured through established methods outlined by the NIH Treatment Fidelity Workgroup on consistency in dose, providers, delivery, receipt and enactment of the intervention. Consultants, Drs. Marazita and Kozikowski will assure fidelity through maintenance of the protocol and its delivery. If questions or concerns arise regarding protocol fidelity, the respective expert will be consulted for assistance and advice. *Dose Consistency*. Initially all patients randomized to intervention groups will have four weeks of either reflexology or meditative practices with their caregiver. Weekly sessions for each of the two therapies will be approximately 45-60 minutes long. Symptom data from the first four weeks will then be evaluated to determine which therapy the dyads will continue with through week 8. *Provider Consistency*. All study providers will pass a demonstration of > 90% proficiency as judged by

the trainers' score on the checklist for both therapies before beginning with caregivers. Caregivers must also achieve 90% accuracy. *Delivery Consistency*. There will be a QA check and booster session conducted biannually for each study provider (those who teach caregivers one or both therapies), with a 90% proficiency in delivery of the therapies. Caregivers are taught and evaluated during intervention weeks 1 and 2. If taught the second therapy after week 4, training and evaluation occurs again at weeks 5 and 6. *Receipt and Enactment Consistency*. The caregiver will also be called by the Education Coordinator every seven days and asked the number of completed sessions since the last weekly call seven days ago. A minimum of 1 session is required, but the exact number of sessions reported by the caregiver will be recorded weekly. Thus, fidelity of the receipt and enactment of each therapy will be documented weekly over the 8-week intervention period.

<u>7e. Incentives.</u> All participants will be mailed a thank-you letter and a local complementary therapy directory after the week 12 data collection. Control caregivers will be offered a complimentary training session of their choice (reflexology or meditative practices). This therapy-based incentive has worked well in the past. 132,152

### 8. Data Collection

<u>8a. Interviews</u>. All patients and caregivers in intervention and control groups will have data collected twice via telephone interviews: baseline and study week 12 to capture post-intervention effects. Study measures have published evidence of reliability and validity with samples of cancer patients and caregivers. The interviews will take 30-45 minutes. If a participant becomes fatigued, we will divide the telephone interview into two phone calls within the same week.

<u>8b. Interviewer Training</u>. The interviewers will call both members of the dyad at intake and week 12. Interviewers will be blinded to the dyad's group assignments. The Education Coordinator will train interviewers via didactic information, written steps, role-playing for difficult interview questions, and return-demonstrations based on our study-specific criteria. In addition, 10% of all interviews will be recorded for QA.

<u>8c. Weekly Calls to Patients.</u> The interviewers will make the weekly calls to all patients to assess symptoms using MDASI (fatigue included) during the 8-week intervention period or an equivalent time frame for the control group. Therefore the attention of asking patients about their symptoms will be equalized across groups. When a symptom is rated at a 7 or higher on the 0-10 scale, patients will be asked to contact their oncology office. For patients randomized to reflexology or meditative practices, weeks 1-4 call data will be used to assess response on fatigue (see definition of symptom response below). If response is not achieved; the patient and caregiver will be re-randomized and weekly calls will continue for weeks 5-8 in the intervention and control groups. The weekly calls will provide documentation of the process of change in symptoms.

<u>8d. Weekly calls to Caregivers</u>. Each intervention caregiver will be called by the Education Coordinator every 7 days to assess the number of sessions conducted with the patient since the last call 7 days ago, as described under Fidelity (section 7b). During weeks 5-8, if rerandomized to add another therapy, the number of sessions will be recorded for the initial and added therapies. The Education Coordinator will make these calls because interviewers need to be blinded to dyad's group assignments.



# 9. Measures of Primary Symptom Outcome - Fatigue

<u>9a. Brief Fatigue Inventory (BFI)</u> <sup>153</sup> (Patients; baseline & week 12). Physical and emotional components of fatigue will be measured with the Brief Fatigue Inventory for rapid assessment of fatigue severity and interference with daily life. The instrument consists of nine items. The first

| Table 3: Measures | | | |
|---|---|---|---|
| Patient Measures | Week | Week<br>12 | Weekly<br>calls |
| T unon mousures | 1 | | |
| 1.a Primary Outcome | | | |
| Physical and Emotional Fatigue (Brief Fatigue Inventory) | Х | Х | |
| Cognitive Fatigue (Attentional Function Index) | Х | Х | |
| 1.b Secondary Outcomes | | | |
| MDASI minus fatigue to avoid redundancy with BFI | Х | Х | |
| PROMIS Depression & Anxiety SF 4 | Х | Х | |
| 1.c Weekly Calls | | | |
| MDASI with fatigue, since no BFI or AFI in brief weekly calls | | | Х |
| 2. Potential Covariates | | | |
| Patient Demographics | Х | | |
| Bayliss Tool (Chronic Conditions) | Х | | |
| Medical Chart: Symptoms & Conditions | | Х | |
| Complementary Therapy Expectancy Scale | Х | | |
| Complementary Therapy Utilization | Х | Х | |
| Satisfaction with Caregiver Involvement Survey | | Х | |
| Caregiver Measures | | | |
| 1. Potential Covariates | | | |
| PROMIS Profile 29 | Х | Х | |
| Caregiver Demographics | Х | | |
| Caregiver Reaction Assessment Tool | Х | Х | |
| Complementary Therapy Expectancy Scale | Х | | |
| Number of Weekly Sessions Completed | | | Х |

three items ask respondents to rate the severity of fatigue "right now," at its "usual" level during the past 24 hours and at its "worst" level during the past 24 hours. Answer choices are on a scale of 0 to 10, where 0=no fatigue and 10=as bad as you can imagine. The remaining six items assess how fatigue affected the following during the past 24 hours: general activity, mood, walking ability, normal work (including work outside the home and daily chores), relations with other people, and enjoyment of life. Responses are on a 0 to 10 scale where 0=does not interfere and 10=completely interferes. Alpha coefficients exceeded .95.

9b. Attentional Function Index (AFI) (Patients; baseline & week 12). 154 The cognitive component of fatigue will be assessed with the 13-item AFI which measures perceived effectiveness in essential daily challenges that require optimal cognition, and has shown consistent reliability in adults with breast cancer. 154,155 In our previous studies with lung cancer, alpha reliabilities were .89 and .91 respectively. 156

# 10. Measures of Secondary Symptom Outcomes.

10a. Symptom Inventory (Patients;

baseline & week 12 & weekly calls). The expanded M.D. Anderson Symptom Inventory (MDASI) evaluates severity of 19 symptoms experienced by cancer patients (i.e., fatigue, pain, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, decreased appetite, drowsiness, dry mouth, sadness, vomiting, numbness/tingling, diarrhea, constipation, sore mouth, rash, hair loss, and cough, and the interference of these symptoms with daily life on the scale from 0=symptom not present to 10=worst imaginable. This instrument has established evidence of reliability and validity in samples of cancer patients. It has been recently updated to include the most common symptoms experienced by patients undergoing modern cancer

treatments.<sup>25</sup> A **single summed** symptom severity score across 18 symptoms (without fatigue, since it is measured in more detail by the BFI and AFI as described in item 9 above) will be used as a secondary outcome in study Aims 1-4 and in building optimal decision rules in exploratory Aim 5.

- 10b. & c. Measures of Secondary Outcomes of Depression and Anxiety. PROMIS-short forms 4: depression and anxiety (Patients; baseline and week 12). 159-162 These two symptoms are not directly covered by MDASI, which includes related items of distress and sadness. Therefore, we include the additional PROMIS measures for these symptoms. PROMIS measures were developed using sophisticated measurement techniques, including Item Response Theory (IRT). 159,163 Testing in more than 21,000 individuals from the U.S. general population has resulted in individual item calibrations that produce t-scores for the general population. The available short forms have evidence of reliability and validity, and have high correlations with IRT-derived scores obtained from extensive item banks. We chose 4-item short forms to minimize respondent burden while maintaining measurement precision.
- 11. Determination of Response on Fatigue during Weeks 1-4 for the Purpose of Rerandomization (Patient; weekly calls). Fatigue response will be assessed based on the fatigue item from MDASI administered in weekly calls to patients. First, we define symptom onset as the date of the weekly call when a symptom for the first time is reported by the patient as moderate or severe according to established and validated cut-points. The cut-points mark the places on a 1-10 severity scale where largest increases in symptom interference occur as severity increases between successive integers ranging from 1 to 10. Thus, the cut-points are anchored in symptom interference with patient's lives. For fatigue, the mild category corresponds to a severity score of 1, moderate category corresponds to scores 2-4, and scores of 5-10 fall into the severe category. Note that the cut-off score of 3 or higher in the inclusion criteria means that at intake patients experience fatigue at a moderate or severe level. Patients who started at severe at onset and ended at moderate or mild by the 4 week observation, and patients who started at moderate and ended at mild, will be called **responders** on fatigue. 164 Since responders demonstrate a substantial improvement anchored to fatigue interference with daily life after 4 weeks, they will continue with the intervention for another 4 weeks. Patients who remain at moderate levels or move to severe at week 4 will be classified as nonresponders. 145,165,166 These patients will be re-randomized to either continue with the same therapy, or add the second therapy, in order to rigorously test the value added by the second therapy in Aims 2 and 3.

# 12. Measures of Dyad Characteristics (Potential Covariates)

- <u>12a. Demographics</u> (Dyads; baseline). Demographics include age, education, work, ethnicity, race, religious affiliation, marital status, and relationship between patient and the friend or family caregiver.
- <u>12b. Chronic Conditions</u> (*Patients; baseline*). The Bayliss tool queries the presence of 20 comorbidities.<sup>167</sup>
- <u>12c. Medical Treatment</u> (Patients; eligibility & week 12). Chart data include radiation, surgery, chemotherapy (dose, type, dates received), co-morbidities, cancer stage, and medications (e.g., supportive agents for pain control, nausea, anxiety, or depressive symptoms) corresponding with the time-on-study. In addition, the Common Terminology Criteria for Adverse Events (CTCAE) data will be collected on side effects and toxicities including anemia and neutropenia.

<u>12d. Complementary Therapy Expectancy Scale</u> (Dyads; baseline). This tool has items on logical thinking and feelings related to complementary therapy use.

<u>12e. Complementary Therapy Utilization</u> (Patients; baseline & week 12). Assesses the use of 24 therapies.

<u>12f. Caregiver Reaction Assessment Tool</u> (Caregiver; baseline and week 12).<sup>170</sup> Caregiver burden will be measured with this tool developed and validated with caregivers of patients with chronic conditions. It has 5 subscales: impact on schedule, caregiver's esteem, family support, impact on health, and impact on finances.

<u>12g. PROMIS Profile-29</u> (Caregivers; baseline & week 12). <sup>159,171</sup> The PROMIS profile instruments are a collection of profile short forms, containing items from one of seven primary PROMIS domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and satisfaction with participation in social roles). The PROMIS Profile-29 includes four items from each primary domain plus a single pain intensity rating. The instrument was developed for the general population and is particularly suitable for the assessment of caregiver health, including symptoms and functioning. Since interventions will be delivered by or practiced with the caregivers, caregiver health may influence the optimal decision rules explored in Aim 5.

<u>12h. Patient Satisfaction with Friend or Family Caregiver Involvement</u>. (Patients; week 12).<sup>172</sup> This survey consists of 5 items that query patient satisfaction with their caregiver involvement. Since the week 12 patient survey is unique for the purposes of this study, it has not been validated with other samples previously. Formal psychometric evaluation will be performed during analysis by Co-PI Dr. Sikorskii who has extensive expertise in measurement. <sup>173-176</sup>

### 13. Protocol Integrity Assessments

<u>13a. Therapy Protocol adherence</u> will be evaluated by the number of completed sessions per week. The Education Coordinator will call the caregiver every seven days and fills out a session form at the end of each weekly call which includes adherence and number of completed sessions during the past seven days.

<u>13b. Attrition Data</u> will be documented when it occurs in association with data collection interviews, including being unable to reach the patient or the patient stating she/he wishes to discontinue. The date and reason, when possible, will be documented. Interviewers will make three attempts for each call.

<u>13c. Training Forms</u> for proficiency will be completed at each training and refresher. The trainers for the reflexologist and meditative practices providers will use a scored proficiency checklist to test study providers accuracy initially and at QA checks every 6 months. Study providers will also use the proficiency checklist when training caregivers at weeks 1 & 2 and if a second therapy is added at weeks 5 & 6.

# 14. Analytic Methods

Data management, tracking and analyses. All data for patients will be entered into the secure web-based database that will be accessible to recruiters and interveners at multiple recruitment sites. To maintain security, data will be stored within a server different from the server of web application. Periodic quality assurance checks of the data will be performed. De-identified data will be transferred into SAS 9.4 for analyses.

14a. Baseline Comparisons and Regression Techniques. To check the baseline equivalence of groups created by the first randomization and the equivalence of subgroups created by the second randomization, the outcome values at baseline and potential covariates will be compared using t-tests, chi-square or Fisher's exact tests. The latter variables include recruitment location, age, sex, site and stage of cancer, type of treatment (e.g., chemotherapy and/or radiation, hormonal therapy, targeted therapy), administration of supportive agents, comorbid conditions, relationship to the caregiver, and living arrangements. If systematic differences are discovered, then the appropriate variables will be included as covariates in further analyses. Outliers will be investigated by inspecting the residuals, and models described below will be fit with and without outliers to examine their influence on the results. Two-sided tests of hypotheses stated below will be performed to determine the superiority of one group versus another as created by first and second randomizations.

14b. Attrition Analyses and Handling of Missing Data. We will compare dyadic characteristics of those who drop out between consent and first randomization to those who continue participation. Following the first randomization, attrition analyses will compare those who drop out according to the second randomization. In addition, we will compare characteristics of those who completed the study with those who did not within their designated group to inform the generalizability of findings. The regression techniques described below allow for missing at random (MAR) mechanisms. The regression techniques described below allow for missing at random (NMAR) mechanisms, then models describing missing mechanisms will be considered (e.g., pattern-mixture models). Since NMAR or MAR assumptions are not directly testable, we will employ sensitivity analyses to investigate the robustness of the results under pattern-mixture or other models.

**Primary Analysis** outcomes: severity of fatigue (primary, physical and emotional from BFI, cognitive from AFI), summed severity index of other symptoms (secondary, from MDASI), depression (secondary, from PROMIS), anxiety (secondary, from PROMIS).

Aim 1, part a), relative effectiveness of reflexology and meditative practices.

**Hypothesis 1.** Patients randomized to the reflexology group will report lower severity of fatigue and lower summed severity score from the MD Anderson symptom inventory at weeks 1-4.

This hypothesis will be tested using statistical model #1 that relates the outcome y at weeks 1-4 to the group assignment variable  $x_1$  (reflexology, meditative practices or control), outcome at baseline  $x_2$ , and other covariates (see baseline comparisons). Additional covariates will include variables used in randomization, due to their potential impact on outcomes. If errors are normally distributed, this model will be fit as a linear mixed effects model (LME), which generalizes classical analysis of repeated measures. Generalized linear mixed effects (GLME) modeling will be used with the appropriate link function and error distribution (e.g., gamma) if the symptom severity outcome is not normally distributed and cannot be normalized using transformations. We are primarily interested in the additive effect of the group variable, and differences in the least square (LS) means will be tested according to the levels of variable  $x_1$ .

**Aim 1, part b),** characteristics of responders and non-responders. Patients who are responders or non-responders on fatigue will be defined as described in measures. The characteristics of

responders and their caregivers will be compared to those of non-responders using t-tests, chisquare or Fisher's exact tests.

**Aim 2, Hypothesis 2.** Patients who do not respond to reflexology on fatigue during weeks 1-4 (1<sup>st</sup> intervention stage) and have the meditative practices added during weeks 5-8 (2<sup>nd</sup> intervention stage), will report lower severity of fatigue and improved 3 secondary outcomes: summed severity index of other symptoms, depression and anxiety, as compared to those who are re-randomized to continue with reflexology alone.

The analytic strategy described under the analyses for Aim 1 will be implemented for the comparison of two groups created by the second randomization. The repeated severity measures during weeks 5-8 and week 12 will be related to study group (reflexology alone versus reflexology and meditative practices), symptom severity during week 4, and covariates (see preliminary analyses). The test of the significance of the coefficient for the group variable will yield a formal test of Hypothesis 2 for the severity of fatigue and other symptoms. PROMIS measures of depression and anxiety obtained in the week 12 interview will be analyzed using general or generalized linear models, and the test of Hypothesis 2 for these 2 secondary outcomes will come from the significance of the coefficient for group assignment in the second randomization.

**Aim 3**, **Hypothesis 3**. Patients who do not respond to meditative practices on fatigue during the weeks 1-4 (1<sup>st</sup> intervention stage) and have the reflexology added during the 2nd intervention stage (weeks 5-8), will report lower severity of fatigue and improved 3 secondary outcomes: summed severity index of other symptoms, depression and anxiety as compared to those rerandomized to continue with meditative practices alone.

The analysis for this aim is the same as the analysis for Aim 2, but will be performed among those who did not respond to meditative practices during weeks 1-4.

**Aim 4, Hypothesis 4:** Patients randomized to intervention sequences beginning with reflexology or meditative practices will report lower severity of fatigue and improved 3 secondary outcomes: summed severity of other symptoms at weeks 1-8 and week 12, depression and anxiety at week 12 compared to controls.

The LME model described under analysis for Aim 1 will be extended to include 8 repeated measures of symptom severity (from weekly calls) and an additional measure from week 12 interview. The test of significance of the explanatory variable reflecting the results of the first randomization will yield a formal test of Hypothesis 4. PROMIS depression and anxiety measures from week 12 interview will be analyzed using generalized linear models with the following explanatory variables: group assignment at first randomization, depression or anxiety (respectively) at baseline, and balancing variables from randomization.

# **Exploratory Analysis: Aim 5.**

To explore which dyadic characteristics observed during weeks 1-4 are associated with optimal patient symptom outcomes at weeks 5-8 and week 12, so as to determine additional tailoring variables for the decision rules of selecting the first intervention stage and switching from the first intervention stage to the second.

The analyses for this aim will help build optimal intervention sequences by determining the optimal decision rule  $(d_1, d_2)$  specifying best first and second intervention stage. This determination is not as simple as determining the best intervention at each stage ignoring future interventions. Such simplistic approaches would ignore longer-term effects of the intervention which was inferior at stage 1, but produced better outcomes in a longer term if simply continued versus combined with another intervention. The analysis approach to this aim therefore follows the maximization method called Q-learning. 167,180-182 The Q-learning algorithm proceeds from right to left in Figure 1, i.e. backwards from the last decision to the first. Two Q-functions will be considered. The function  $Q_2(H_2) = E[Y_2|H_2]$  is the expectation of the second stage outcome  $Y_2$ given history after 2 stages, denoted by  $H_2$ : dyadic characteristics, outcomes observed during weeks 1-8 and week 12, and interventions received. The function  $Q_1(H_1) = E[Y_1 + \max Q_2(H_2)]$ uses history through the first intervention stage H<sub>1</sub>. The conditional expectations in the Qfunctions will be estimated from regression analyses for the outcomes of severity of fatigue. summed severity of other symptoms, depression & anxiety, and the optimal decision rule will be found using backward induction by maximizing these functions. 183,184 Due to caregiver involvement in intervention delivery, caregiver characteristics including measures of symptoms (described in the measures section) will be explored, as the optimal decision rules may be based on both patient and caregiver factors. The Q-learning method will be implemented in SAS PROC QLEARN<sup>129</sup> developed by Murphy and colleagues. <sup>185</sup> The procedure uses a generalization of Q-learning, which allows treatments and covariates to vary over time, a feature especially relevant to this trial that has weekly symptom assessments. Using this procedure, we will identify tailoring variables that can be used to operationalize the decision rules of selecting the first intervention and switching from the first intervention stage to the second. These decision rules can then undergo testing in a future confirmatory RCT.

# 15. Potential Difficulties/Limitations and Alternative Approaches

Since randomizations may not account for all possible error sources, we will adjust for baseline values of outcomes in the analysis to provide added control over possible confounding pre-intervention influences. One primary (fatigue), 3 secondary outcomes (summed severity of other symptoms, depression & anxiety) and the hypotheses are all stated a priori. In the exploratory analyses, the issue of multiple testing will be addressed by employing the Benjamini-Hochberg or Hochberg adjustment to control for the false discovery rate. Because multiplicity adjustments are controversial, all results will be presented both adjusted and unadjusted.

| Table 4. Timeline | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Months | 1-6 | 7-12 | 13-18 | 19-24 | 25-30 | 31-36 | 37-42 | 43-48 |
| Contracts, site IRBs, manuals, training, database programming | Х | | | | | | | |
| Enrollment, interviews, interventions, medical record audits | | Х | Х | Х | Х | Х | Х | |
| Conduct QA, data safety and attrition monitoring | | Х | Х | Х | Х | Х | Х | |
| Set up for analysis, conduct analysis, report | | Х | | Х | | Х | | Х |

# 16. Data Sharing

Findings from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings.

# **Literature Cited**

- **1.** ASCO Report. The state of cancer care in America, 2014: a report by the American Society of Clinical Oncology. *Journal of Oncology*. 2014:1-25.
- **2.** Butt Z, Rosenbloom SK, Abernethy AP, et al. Fatigue is the most important symptom for advanced cancer patients who have had chemotherapy. *Journal of the National Comprehensive Cancer Network.* 2008;6(5):448-455.
- **3.** Grabsch B, Clarke DM, Love a, et al. Psychological morbidity and quality of life in women with advanced breast cancer: A cross-sectional survey. *Palliative and Supportive Care*. 2006;4:47-56.
- **4.** National Cancer Institute. About Cancer Survivorship Research: Survivorship Definitions. 2009; <a href="http://cancercontrol.cancer.gov/ocs/definitions.html">http://cancercontrol.cancer.gov/ocs/definitions.html</a>. Accessed Feb. 27, 2009.
- **5.** Wyatt G, Sikorskii A, Rahbar M, Victorson D, You M. Health-related quality of life outcomes: A reflexology trial with patients with advanced-stage breast cancer. *Oncology Nursing Forum*. November 2012;39(6):568-577.
- **6.** Wyatt G, Sikorskii A, Tamkus D, You M. Quality of life among advanced breast cancer patients with and without distant metastasis. *European Journal of Cancer Care*. 2013;22:272-280.
- **7.** Reyes-Gibby C, Anderson KO, Morrow PK, Shete S, Hassan S. Depressive symptoms and health-related quality of life in breast cancer survivors. *Journal of Womens Health*. 2012;21(3):311-318.
- **8.** Jeffe DB, Perez M, Luiu Y, Collins KK, Aft RL, Schootman M. Quality of life over time in women diagnosed with ductal carcinoma in situ, early-stage invasive breast cancer, and age-matched controls. *Breast Cancer Research and Treatment*. 2012;134(1):379-391.
- **9.** Aranda S, Schofield P, Weih L, et al. Mapping the quality of life and unmet needs of urban women with metastatic breast cancer. *European Journal of Cancer Care*. 2005;14(3):211-222.
- **10.** Barsevick AM, Cleeland CS, Manning DC, et al. ASCPRO Recommendations for the Assessment of Fatigue as an Outcome in Clinical Trials. *J Pain Symptom Manage*. 2010;39(6).
- **11.** Kroenke K. Studying symptoms: sampling and measurement issues. *Ann Intern Med.* May 1 2001;134(9 Pt 2):844-853.
- **12.** Armes J. The experience of cancer-related fatigue. *Fatigue in Cancer.* 2004.

- **13.** Higginson IJ, Armes J, Krishnasarny M. Fatigue in Cancer: Introduction. *Oxford University Press*. 2004:xvii-xxi.
- **14.** Lehto R, Wyatt G. Perceptions about Using Mindfulness Therapy: A Lung Cancer Focus Group Study. *Cancer Nursing: An international Journal for Cancer Care.* 2013:E51-60.
- **15.** Cella D, Lai J, Chang C, Peterman A, Slavin M. Fatigue in cancer patients compared with fatigue in the general United States population. *Cancer.* 2002;94(2):528-538.
- **16.** Piper B, Dibble S, Dodd M, Slaughter R, Paul S. The revised Piper Fatigue Scale: Psychometric evaluation in women with breast cancer. *Oncology Nursing Forum*. 1998;25(4):677-684.
- **17.** Mitchell S, Bergre A. Cancer-related fatigue: the evidence base for assessment and management. *Cancer*. 2006;12(5):374-387.
- **18.** Nail L. Fatigue in patients with cancer. *Oncol Nurs Forum.* 2002;29(3):537.
- **19.** Huang H, Chen M, Liang J, Miaskowski C. Changes in and predictors of severity of fatigue in women with breast cancer: A longitudial study. *International Journal of Nursing Studies*. 2014;51:582-592.
- **20.** Choi J, Tate J, Hoffman L, et al. Fatigue in Family Caregivers of Adult Intensive Care Unit Survivors. *Journal of Pain and Symptom Management*. 2014;48(3):353-363.
- 21. Schrepf A, Clevenger L, Christensen D, et al. Cortisol and inflammatory processes in ovarian cancer patients following primary treatment: relationships with depression, fatigue, and disability. *Brain Behav Immun*. Mar 2013;30 Suppl:S126-134.
- **22.** Clevenger L, Schrepf A, Christensen D, et al. Sleep disturbance, cytokines, and fatigue in women with ovarian cancer. *Brain Behav Immun*. Oct 2012;26(7):1037-1044.
- **23.** Bower JE, Ganz PA, Irwin MR, Kwan L, Breen EC, Cole SW. Inflammation and behavioral symptoms after breast cancer treatment: Do fatigue, depression and sleep disturbance share a common underlying mechanism? . *Journal of Clinical Oncology.* 2011;29(26):3517-3522.
- **24.** Gift A, Jablonski A, Stommel M, Given C. Symptom clusters in elderly patients with lung cancer. *Oncol Nurs Forum.* 2004;31(2):203-209.
- **25.** Cleeland CS, Fengmin Z, Chang VT, et al. The symptom burden of cancer: Evidence for a core set of cancer-related and treatment-related symptoms from the eastern cooperative oncology group symptom outcomes and practice patterns study. *Cancer* 2013.
- 26. Mendoza TR WX, Lu C, Palos GR, Liao, Z, Mobley GM, Kapoor S, Cleeland CS. Measuring the symptom burden of lung cancer the validity and utility of the lung cancer module of the M.D. Anderson Symptom Inventory. *Oncologist*. 2011;16(2):217-227.
- **27.** Henoch I, Bergman B, & Danielson E. Dyspnea experience and management strategies in patients with lung cancer. *Psycho-Oncology*. 2008;17: 709-715.
- **28.** Zhao I, & Yates P. Non-pharmacological interventions for breathlessness management in patients with lung cancer: a systematic review. *Palliative medicine*. 2008;22:693-701.

- **29.** Lehto RH, Wyatt G, Sikorskii A, Tesnjak I, Kaufman VH. Home-based Mindfulness Therapy for Lung Cancer Symptom Management: A Randomized Feasibility Trial. *Psycho-oncology*. 2015.
- **30.** Zabora J, Brintzenhofesoc K, Curbow B, Hooker C, S P. The prevalence of psychological distress by cancer site. *Psycho-Oncology*. 2001;10:19-28.
- **31.** Wurtzen H, Dalton SO, Elsass P, et al. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. *Eur J Cancer*. Apr 2013;49(6):1365-1373.
- **32.** Lehto R. Mindfulness Therapy for Individuals with Lung Cancer. Vol GA013811CTSIL: Michigan State University, Clinical Translational & Science Institute.
- **33.** Wyatt G, Sikorskii A, Holmstrom A, Luo Z. Home Based Symptom Management via Reflexology for Advanced Breast Cancer Patients *National Institutes of Health, National Cancer Institute grant # R01CA157459-01.* 2011-2016.
- **34.** Tacón AM, Caldera YM, Ronaghan C. Mindfulness-based stress reduction in women with breast cancer. . *Families Systems & Health*. 2004;22:193-203.
- **35.** Carlson LE, Speca M, Patel KD, & Goodey E. Mindfulness-based stress reduction in relation to quality of life,mood, symptoms of stress and levels of cortisone, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. *Psychoneuroendocrinology.* 2004;29:448-474.
- **36.** Van der Lee M, & Garssen B. Mindfulness-based cognitive therapy reduces chronic cancer-related fatigue: a treatment study. *Psycho-Oncol.* 2012;21:264-272.
- **37.** Sarna L, Evangelista L, Tashkin D, et al. Impact of respiratory symptoms and pulmonary function on quality of life of long-term survivors of non-small cell lung cancer. *Chest.* 2004;125:439-446.
- **38.** Stenberg U, Ruland CM, Miaskowski C. Review of the literature on the effects of caring for a patient with cancer. *Psychooncology*. 2010;19:1013-1025.
- **39.** American Cancer Society. Family Caregivers. 2011; <a href="http://www.cancer.org/Research/ResearchProgramsFunding/BehavioralResearchCenter/WhatthebehavioralResearchCenterDoes/family-caregivers">http://www.cancer.org/Research/ResearchProgramsFunding/BehavioralResearchCenter/WhatthebehavioralResearchCenterDoes/family-caregivers</a>. Accessed October 10, 2012.
- **40.** Newcott B. The Silent cry of the caregiver. *AARP Magazine*. Vol 55. Washington DC: AARP; 2012:86-91.
- **41.** National Alliance for Caregiving & AARP. *Caregiving in the U.S.* Washington D.C.2004.
- **42.** National Family Caregivers Association, Family Caregiver Alliance. *Prevalence, Hours and Economic Value of Family Caregiving, Updated State-by-State Analysis of 2004 National Estimates (by Peter S. Arno, PhD).* Kensington, MD: NFCA & San Francisco, CA: FCA2006.
- **43.** Arno PS. Economic Value of Informal Caregiving: 2004. 2006; <a href="http://www.va.gov/occ/Conferences/caregiverforum/Docs/Arno-Handout.pdf">http://www.va.gov/occ/Conferences/caregiverforum/Docs/Arno-Handout.pdf</a>.

- Bevans M, Sternberg E. Caregiving burden, stress, and health effects among family caregivers of adult cancer patients. *JAMA*. 2012;37(4):398-403.
- **45.** Bultz BD, Speca M, Brasher PM, Geggie PH, Page SA. A randomized controlled trial of a brief psychoeducational support group for partners of early stage breast cancer patients. *Psychooncology*. 2000;9(4):303-313.
- **46.** Carlson LE, Ottenbreit N, St Pierre M, Bultz BD. Partner understanding of the breast and prostate cancer experience. *Cancer Nursing*. 2001;24(3):231-239.
- **47.** Given B, Given C, Sikorskii A, Jeon S, Sherwood P, Rahbar M. The impact of providing symptom management assistance on caregiver reaction: Results of a randomized trial. *Journal of Pain and Symptom Management*. 2006;32(5):433-443.
- **48.** Given B, Sikorskii A, Given C, You M. Effects of assisting cancer patients with symptom management on fmaily members reports of burden and depression. *Psychooncology*. 2009;18(Suppl 2):S70-S71.
- **49.** Kozachik S, Wyatt GK, Given CW, Given B. Patterns of Use of Complementary Therapies Among Cancer Patients and Their Family Caregivers. *Cancer Nursing*. 2006;29(2):84-94.
- **50.** Cantarero-Villanueva I, Fernandez-Lao C, Cuesta-Vargas A, Moral-Avila R, Fernandez-de-las-Penax C, Arroyo-Morales M. The Effectiveness of a Deep Water Aquatic Exercise Program in Cancer-Related Fatigue in Breast Cancer Survivors: A Randomized Controlled Trial. *Archives of Physical Medicine and Rehabilitation*. 2013;94:221-230.
- **51.** Bower JE, Garet D, Sternlieb B, et al. Yoga for persistent fatigue in breast cancer survivors: a randomized controlled trial. *Cancer.* Aug 1 2012;118(15):3766-3775.
- **52.** Velthuis MJ, Agasi-Idenburg SC, Aufdemkampe G, Wittink HM. The Effect of Physical Exercise on Cancer-related Fatigue during Cancer Treatment: a Meta-analysis of Randomised Controlled Trials. *Clinical Oncology.* 2010;22:208-221.
- Dodd M, Cho M, Miaskowski C, et al. A Randomized Controlled Trial of Home-Based Exercise for Cancer-Related Fatigue in Women During and After Chemotherapy With or Without Radiation Therapy. *Cancer Nursing*. 2012;33(4):245-257.
- **54.** Hawkes AL, Chambers SK, Pakenham KI, et al. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. *J Clin Oncol.* 2013;31(18):2313-2321.
- **55.** Kim S, Shin MS, Lee H, et al. Randomized Pilot Test of a Simultaneous Stage-Matched Exercise and Diet Intervention for Breast Cancer Survivors. *Oncol Nurs Forum*. 2011;38(2):97-106.
- **56.** Bourke L, Gilbert S, Hooper R, et al. Lifestyle Chances for Improving Disease-specific Quality of Life in Sedentary Men on Long-term Androgen-Deprivation Therapy for Advanced Prostate Cancer: A Randomised Controlled Trial. *European Urology*. 2014;65:865-872.

- **57.** Bourke L, Doll H, Crank H, Daley A, Rosario D, Saxton J. Lifestyle Intervention in Men with Advanced Prostate Cancer Receiving Androgen Suppression Therapy: A Feasibility Study. *Cancer Epidemiol Biomarkers Prev.* 2011;20(4):647-657.
- **58.** Bourke L, Thompson G, Gibson D, et al. Pragmatic Lifestyle Intervention in Patients Recovering From Colon Cancer: A Randomized Controlled Pilot Study. *Arch Phys Med Rehabil.* 2011;92:749-755.
- **59.** Wyatt G, Sikorskii A, Wills CE, Ahn HS. Complementary and alternative medicine use, spending, and quality of life in early stage breast cancer. . *Nursing Research*. 2010;59(1):58-66.
- **60.** Lowry SJ, Loggers ET, Bowles EJ, Wagner EH. Evidence gaps in advanced cancer care: community-based clinicians' perspectives and priorities for comparative effectiveness research. *J Oncol Pract.* 2012;8(3 Suppl).
- **61.** Lyman GH. Comparative effectiveness research in oncology. *Oncologist.* 2013;18(6):752-759.
- Boon HS, Olatunde F, Zick SM. Trends in complementary/alternative medicine use by breast cancer survivors: Comparing survey data from 1998 and 2005. *BMC Womens Health* 2007; <a href="http://www.biomedcentral.com/content/pdf/1472-6874-7-4.pdf">http://www.biomedcentral.com/content/pdf/1472-6874-7-4.pdf</a>, 7(4).
- **63.** Grady PA. Translational research and nursing science. *Nurs Outlook*. May-Jun 2010;58(3):164-166.
- **64.** Eisenberg D, Davis R, Ettner S, Appel S, Rompany M, Kessler R. Trends in alternative medicine uses in the United States, 1990-1997. *Journal of the American Medical Association*. 1998;280(18):1569-1575.
- National Health Interview Survey. Percentage of Adults Aged >18 Years Who Used Complementary and Alternative Medicine (CAM), by Selected Diseases and Conditions and Sex. 2008; <a href="http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5735a5.htm">http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5735a5.htm</a>. Accessed November 5, 2012.
- 66. Morano C, Giunta N, Parikh N, Panuska S, Fahs M, Gallo W. Mind-Body Techniques, Race-Ethnicity, and Depression among Urban Senior Center Participants. *Health & Social Work*. 2013;38(3):167-172.
- **67.** Lee M, Lin S, Wrensch M, Adler S, Eisenberg D. Alternative Therapies Used by Women with Breast Cancer in Four Ethnic Populations. *Journal of the National Cancer Institute*. 2000;92(1):42-47.
- **68.** Villa-Caballero L, Morello C, Chynoweth M, et al. Ethnic differences in complimentary and alternative medicine use among patients with diabetes. *Complementary Therapies in Medicine*. 2010;18:241-248.
- 69. Neiberg RH, Aickin M, Grzywacz JG, et al. Occurrence and co-occurrence of types of complementary and alternative medicine use by age, gender, ethnicity, and education among adults in the United States: The 2002 National Health Interview Survey. *Journal of Alternative & Complementary Medicine*. 2011;17(4):363-370.

- 70. Seburg E, Horvath K, Garwick A, McMorris B, Vehe R, Scal P. Complementary and Alternative Medicine Use Among Youth With Juvenile Arthritis: Are Youth Using CAM, But Not Talking About It? *Journal of Adolescent Health*. 2012;51:200-202.
- 71. Fries C. Ethincity and the use of "accepted" and "rejected" complementary/alternative medical therapies in Canada: evidence from the Canadian Community Health Survey. *Issues in Health and Health Care Related to Race/Ethnicity, Immigration, SES and Gender Research in the Sociology of Health Care.* 2012;30:113-131.
- **72.** National Institutes of Health, National Center for Complementary and Alternative Medicine. What is CAM? 2014; <a href="http://nccam.nih.gov/health/whatiscam/">http://nccam.nih.gov/health/whatiscam/</a>.
- **73.** Deng G, Cassileth B. Complementary or alternative medicine in cancer care- myths and realities. *Nature Reviews Clinical Oncology.* 2013;10:656-664.
- **74.** Stephenson N, Swanson M, Dalton J, Keefe FJ, Engelke M. Partner-delivered reflexology: Effects on cancer pain and anxiety. *Oncology Nursing Forum.* 2007;34(1):127-132.
- **75.** Foley E, Baillie A, Huxter M, Price M, & Sinclair E. Mindfulness-based cognitive therapy for individuals whose lives have been affected by cancer: A randomized controlled trial. *Journal of Consulting and Clinical Psychology.* 2010;78:72-79.
- **76.** Watson S, Voner V. *Practical Reflexology: Interpretation and Techniques*: McGraw-Hill Companies, Incorporated; 2008.
- **77.** Ernst E. Is reflexology an effective intervention: A systematic review of randomized controlled trials. *Medical Journal of Australia*. 2009;191(5):263.
- **78.** Stephenson N, Weinrich S, Tavakoli A. The effects of foot reflexology on anxiety and pain inpatients with breast and lung cancer. *Oncol Nurs Forum.* 2000;27:67-72.
- **79.** Hodgson H. Does reflexology impact on cancer patients' quality of life? *Nurs Stand.* 2000;14(31):33-38.
- **80.** Wilkinson S, Lockhart K, Gambles M, Storey L. Reflexology for symptom relief in patients with cancer. *Cancer Nursing*. 2008;Sept-Oct(5):354-360.
- **81.** Quattrin R, Zanini A, Buchini S, et al. Use of reflexology foot massage to reduce anxiety in hospitalized cancer patients in chemotherapy treatment: Methodology and outcomes. *Journal of Nursing Management*. 2006;14(2):96-105.
- **82.** Stephenson N, Dalton JA, Carlson J. The effect of foot reflexology on pain in patients with metastatic cancer. *Appl Nurs Res.* 2003;16(4):284-286.
- **83.** Tsay S, Chen H, Chen S, Lin H, Lin K. Effects of reflexotherapy on acute postoperative pain and anxiety among patients with digestive cancer. *Cancer Nursing*. 2008;31(2):109-115.
- **84.** Sharp DM, Walker MB, Chaturvedi A, et al. A randomized, controlled trial of the psychological effects of reflexology in early breast cancer. *Eur J Cancer*. 2010;46(2):312-322.

- **85.** Ernst E, White A. The BBC survey of complementary medicine use in the UK. *Complementary Therapy in Medicine*. 2000;8(1):32-36.
- **86.** Kabat-Zinn J. *Full Catastrophe Living: Using The Wisdom Of Your Body And Mind To Face Stress, Pain, and Illness.* 15 ed. New York: Delta Trade Paperbacks; 2009.
- 87. Branstrom R, Kvillemo P, Brandberg Y, Moskowitz JT. Self-report mindfulness as a mediator of psychological well-being in a stress reduction for cancer patients A randomized study. *Annals of Behavioral Medicine*. 2010;39:151-161.
- **88.** Arch JJ, Craske MG. Mechanisms of mindfulness: Emotion regulation following a focused breathing induction. *Behaviour Research and Therapy.* 2006;44(1849-1858).
- **89.** Tacon AM, Caldera YM, Ronaghan C. Mindfulness-based stress reduction in women with breast cancer. *Families, Systems & Health.* 2004;22:193-203.
- **90.** Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress rediction in relation to quality of life, mood, symptoms of stress and levels of cortisone, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. *Psychoneuroendocrinology*. 2004;29:448-474.
- **91.** Shapiro SF, Carlson LE, Astin JA, Freedman B. Mechanisms of mindfulness. *Journal of Clinical Psychology* 2006;62:373-386.
- **92.** Ledesma D, Kumano H. Mindfulness-based stress reduction and cancer: a meta-analysis. *Psycho-Oncology*. 2009;18:571-579.
- 93. Shennon C, Payne S, & Fenlon D. What is the evidence for the use of mindfulness-based interventions in cancer care? A review. "Psycho-Oncology, ". 2010;18:571-579.
- **94.** Matchim Y, Armer JM, Stewart BR. Mindfulness-based stress reduction among breast cancer survivors: a literature review and discussion. *Oncol Nurs Forum*. Mar 2011;38(2):E61-71.
- **95.** Carlson LE, Speca M, Faris P, Patel KD. One year pre-post intervention follow-up of psychological, immune, endocrine and blood pressure outcomes of mindfulness-based stress reduction (MBSR) in breast and prostate cancer outpatients. *Brain, Behavior and Immunity*. 2007;21:1038-1049.
- **96.** Carlson LE, & Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. *International Journal of Behavioral Medicine*. 2005;12:278-285.
- **97.** Tacón AM, Caldera YM, Ronaghan C. Mindfulness-based stress reduction in women with breast cancer. *Families Systems & Health*. 2004;22(2):193-203.
- **98.** Witek-Janusek L, Albuquerque K, Chroniak KR, Chroniak C, Durazo-Arvizu R, Mathews HL. Effect of mindfulness based stress reduction on immune function, quality of life and coping in women newly diagnosed with early stage breast cancer. *Brain Behav Immun*. Aug 2008;22(6):969-981.

- **99.** Shapiro SL, Bootzin RR, Figueredo AJ, Lopez AM, Schwartz GE. The efficacy of mindfulness-based stress reduction in the treatment of sleep disturbance in women with breast cancer: an exploratory study. *Journal of Psychosomatic Research*. 2003;54:85–91.
- **100.** Monti DA, Peterson C, Kunkel EJ, et al. A randomized, controlled trial of mindfulness-based art therapy (MBAT) for women with cancer. *Psycho-Oncology*. 2006;15:363–373.
- **101.** Lengacher CA, Johnson-Mallard V, Post-White J, et al. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. *Psycho-Oncology*. 2009;18:1261-1272.
- **102.** Lengacher CA, Reich RR, Post-White J, et al. Mindfulness based stress reduction in post-treatment breast cancer patients: an examination of symptoms and symptom clusters. *J Behav Med.* Feb 2012;35(1):86-94.
- **103.** Bränström R, Kvillemo P, Brandberg Y, & Moskowitz JT. Self-report mindfulness as a mediator of psychological well-being in a stress reduction for cancer patients A randomized study. *Annals of Behavioral Medicine*. 2010;39:151-161.
- **104.** Andersen SR, Wurtzen H, Steding-Jessen M, et al. Effect of mindfulness-based stress reduction on sleep quality: results of a randomized trial among Danish breast cancer patients. *Acta Oncol.* Feb 2013;52(2):336-344.
- **105.** Garland SN, Carlson LE, Cook S, Lansdell L, & Speca M. A non-randomized comparison of mindfulness-based stress reduction and healing arts programs for facilitating post-traumatic growth and spirituality in cancer outpatients. *Support Care Cancer*. 2007;15(8):949–961.
- **106.** Matchim Y, Armer JM, Stewart BR. Effects of mindfulness-based stress reduction (MBSR) on health among breast cancer survivors. *West J Nurs Res.* Dec 2011;33(8):996-1016.
- **107.** Monti DA, Kash KM, Kunkel EJ, et al. Changes in cerebral blood flow and anxiety associated with an 8-week mindfulness programme in women with breast cancer. *Stress Health*. Dec 2012;28(5):397-407.
- **108.** Matousek RH, Pruessner JC, Dobkin PL. Changes in the cortisol awakening response (CAR) following participation in mindfulness-based stress reduction in women who completed treatment for breast cancer. *Complement Ther Clin Pract.* May 2011;17(2):65-70.
- **109.** Matousek RH, Dobkin PL. Weathering storms: a cohort study of how participation in a mindfulness-based stress reduction program benefits women after breast cancer treatment. *Curr Oncol.* Aug 2010;17(4):62-70.
- **110.** Henderson VP, Clemow L, Massion AO, Hurley TG, Druker S, Hebert JR. The effects of mindfulness-based stress reduction on psychosocial outcomes and quality of life in early-stage breast cancer patients: a randomized trial. *Breast Cancer Res Treat*. Jan 2012;131(1):99-109.
- **111.** McVicar AJ, Greenwood CR, Fewell F, D'Arcy V, Chandrasekharan S, Alldridge LC. Evaluation of anxiety, salivary cortisol and melatonin secretion following reflexology treatement: A pilot study in healthy individuals. *Complement Ther Clin Pract.* 2007;13(3):137-145.

- Hölzel BK, Carmody J, Vangel M, et al. Mindfulness practice leads to increases in regional brain gray matter density. *Psychiatry Research: Neuroimaging*. 2011;191:36-43.
- **113.** Nahum-Shani I, Qian M, Almirall D, et al. Q-learning: A data analysis method for constructing adaptive interventions. *Psychological methods*. 2012;17(4):478.
- **114.** Nahum-Shani I, Qian M, Almirall D, et al. Experimental design and primary data analysis methods for comparing adaptive interventions. *Psychological methods*. 2012;17(4):457.
- **115.** Kohara H, Miyauchi T, Suehiro Y, Ueoka H, Takeyama H, Morita T. Combined modality treatment of aromatherapy, footsoak, and reflexology relieves fatigue in patients with cancer. *J Palliat Med.* 2004;7(6):791-796.
- **116.** Ong JC, Shapiro SL, & Manber R. Mindfulness meditation and cognitive behavioral therapy for insomnia: A naturalistic 12-month follow-up. *Explore*. 2009;5.
- **117.** Radin D, Stone J, Levine E, et al. Compassionate intention as a therapeutic intervention by partners of cancer patients: Effects of distant intention on the patients' autonomic nervous system. *Explore*.4(4):235-243.
- **118.** Brotto LA, Heiman JR, Goff B. A psychoeducational intervention for sexual dysfunction in women with gynecological cancer. *Arch Sexual Behavior*. 2008;37(2):317-329.
- **119.** Chakraborty B, Murphy S. Inference for non-regular parameters in optimal dynamic treatment regimes. *Statistical Methods in Medical Research*. 2010;19(3):317-343.
- **120.** Collins L, Murphy S, Bierman K. A conceptual framework for adaptive preventive interventions. *Prevention Science*. 2004;5(3):185-196.
- **121.** Rush AJ, Fava M, Wisniewski SR, et al. Sequenced treatment alternatives to relieve depression (STAR\*D): Rationale and design. *Controlled Clinical Trials.* 2003;25(1):119-142.
- **122.** Schneider LS, Tariot PN, Lyketsos CG, et al. National Institute of Mental Health clinical antipsychotic trials of intervention effectiveness (CATIE): Alzheimer disease trial methodology. *American Journal of Geriatric Psychiatry*. 2001;9(4):346-360.
- **123.** Thall PF, Millikan RF, Sung HG. Evaluating multiple treatment courses in clinical trials. *Statistics in Medicine*. 2000;19(8):1011-1128.
- **124.** Wahed AS, Tsiatis AA. Optimal estimator for the survival distribution and related quantities for treatment policies in two-stage randomized designs in clinical trials. *Biometrics*. 2004;60(1):124-133.
- **125.** Collins L, Murphy S, Nair VN, Strecher VJ. A strategy for optimizing and evaluating behavioral interventions. *Annals of Behavioral Medicine*. 2005;30(1):65-73.
- **126.** Given CW, Given B, Azzouz F, Kozachik S, Stommel M. Predictors of pain and fatigue in the year following diagnosis among elderly cancer patients. *Journal of Pain and Symptom Management*. 2001;21(6):456-466.

- **127.** Stanton AL, Bernaards CA, Ganz PA. The BCPT symptom scales: a measure of physical symptoms for women diagnosed with or at risk for breast cancer. *J Natl Cancer Inst.* Mar 16 2005;97(6):448-456.
- **128.** Cooley ME, Short TH, Moriarty HJ. Symptom prevalence, distress, and change over time in adults receiving treatment for lung cancer. *Psychooncology*. Oct-Nov 2003;12(7):694-708.
- **129.** PROC QLEARN (Version 1.0) 2012; <a href="http://methodology.psu.edu/downloads/procqlearn">http://methodology.psu.edu/downloads/procqlearn</a>. Accessed May 5, 2013.
- **130.** Given C, Wyatt G, Given B. A Complementary Therapy Intervention for Supportive Care of Cancer Patients. *West Michigan Cancer Center, Michigan State University, and the Mary Margaret Walther Program.* 1998-2002.
- **131.** Wyatt G, Sikorskii A, Siddiqi A. Feasibility of a reflexology and guided imagery intervention during chemotherapy: Results of a quasi-experimental study. *Oncology Nursing Forum*. 2007;34(3):635-642.
- **132.** Wyatt G, Sikorskii A, Holmstrom A, Luo Z. Home Based Symptom Management via Reflexology for Advanced Breast Cancer Patients: National Institutes of Health, National Cancer Institute grant # R01CA157459-01; 2011-2016.
- **133.** Wyatt G. Complementary and alternative therapy interventions used by cancer patients. . *In:* Given, C., Given, B, Champion, V., Kozachik, s., eds. Evidence Based Behavioral Interventions in Oncology: State of the knowledge across the cancer care continuum. 2003:292-331.
- **134.** Wyatt G, Beckrow K, Gardiner J, Pathak DR. Predictors of post-surgical sub-acute emotional and physical well-being among women with breast cancer. *Cancer Nurs.* 2008;31(2):E28-E39.
- **135.** Wyatt G, Friedman LS, Given C, Given B, & Beckrow K. Complementary therapy use among older cancer patients. *Cancer Practice*. 1999;7:136-144.
- **136.** Wyatt G, Friedman-Donze L. The long-term quality of life (LTQL) instruments for female cancer survivors. In: Strickland O, Dilorio C, eds. *Measurement of Nursing Outcomes: Self Care and Coping.* Vol 3. 2nd ed: Springer Publishing Company; 2003:216-226.
- **137.** Wyatt G, Given B, & Given C. A subacute care intervention for short-stay breast cancer surgery: U.S. Army Medical Research. *Department of Defense*. 1996-2001.
- **138.** Wyatt G, Kurtz ME, Liken M. Breast Cancer Survivors: An exploration on quality of life issues. *Cancer Nurs.* 1993;16(6):440-448.
- **139.** Wyatt G, L.F. D, & Beckrow K. Efficacy of an In-home Nursing Intervention Following Short-stay Breast Cancer Surgery. *Research in Nursing & Health.* 2004;27:322-331.
- **140.** Wyatt G, Sikorskii A, Bush TR, Mukherjee R. Team Science of Nursing, Engineering, Statistics, and Practitioner in the Development of a Robotic Reflexology Device. *Journal of the Society for Integrative Oncology.* 2010;8(1):14-19.
- **141.** Wyatt G, Sikorskii A, Rahbar MH, Victorson D, Adams L. Intervention fidelity: Aspects of Complementary and Alternative Medicine (CAM) research. *Cancer Nursing*. 2010;33(5):331-342.

- **142.** Wyatt GK, & Post-White J. Future direction of complementary and alternative medicine (CAM) education and research. *Seminars in Oncology Nursing*. 2005;21:215-224.
- **143.** Sikorskii A, Given CW, You M, Jeon S, Given BA. Response analysis for multiple symptoms revealed differences between arms of a symptom management trial. *Journal of Clinical Epidemiology*. 2009;62(7):716-724.
- **144.** Sikorskii A, Given CW, Given B, et al. Symptom management for cancer patients: a trial comparing two multimodal interventions. *J Pain Symptom Manage*. Sep 2007;34(3):253-264.
- **145.** Given B, Given C, Sikorskii A, et al. Establishing mild, moderate and severe scores for cancer related symptoms: How consistent and clinically meaningful are interference based severity cut points? *Journal of Pain and Symptom Management*. 2008;35(2):126-135.
- **146.** Jeon S, Given C, Sikorskii A. The utility of screening in the design of trials for symptom management in cancer. *Journal of Pain and Symptom Management*. 2009;38(4):606-614.
- **147.** Sikorskii A, Given C, Given B, Jeon S, Decker V, Decker D. Symptom management for cancer patients: A trial comparing two multimodal interventions. *Journal of Pain and Symptom Management*. 2007;34(3):253-264.
- **148.** Sikorskii A, Wyatt GK, Siddiqi A, Tamkus D. Recruitment and retention of women with advanced breast cancer in a complementary and alternative medicine (CAM) trial. *Evid Based Complement Alternat Med.* 2009:Doi: 10.1093/ecam/nep1051.
- **149.** Taves DR. Minimization: a new method of assigning patients to treatment and control groups. *Clin Pharmacol Ther.* May 1974;15(5):443-453.
- **150.** National Center for Complementary and Alternative Medicine. NIH NCCAM Congressional Justification 2012. 2012. Accessed June 19, 2013.
- **151.** Bellg AJ, Borrelli B, Resnick B, et al. Enhancing Treatment Fidelity in Health Behavior Change Studies: Best Practices and Recommendations From the NIH Behavior Change Consortium. *Health Psychol.* 2004;23(5):443-451.
- **152.** Wyatt G, Sikorskii A, Rahbar MH. Reflexology: An Intervention for Advanced Breast Cancer: NIH/NCI; 2005-2011.
- **153.** Mendoza T, Wang S, Cleeland CS, et al. The rapid assessment of fatigue severity in cancer patients. *Cancer*. 1999;85(5):1186-1196.
- **154.** Cimprich B. The Attentional Function Index-a self-report cognitive measure. *Psycho-oncology.* 2010; published online in Wiley InterScience: 9.
- **155.** Cimprich B. Attentional fatigue following breast cancer surgery. *Research in Nursing & Health.* 1992;15:199-207.
- **156.** Lehto RH. Pre- and Post-operative Self-reported Cognitive Effectiveness and Worry in Patients with Suspected Lung Malignancy. *Oncology Nursing Forum.* 2013;40(3):e135-141.

- **157.** Cleeland CS. Symptom burden: Multiple symptoms and their impact as patient-reported outcomes. *Journal of the National Cancer Institute Monographs*. 2007;37:16-21.
- **158.** Cleeland CS, Mendoza T, Wang XS, Chou C, Harle MT, Engstrom MC. Assessing symptom distress in cancer patients: The M.D. Anderson symptom inventory. *Cancer*. 2000;89(7):1634-1646.
- **159.** Cella D, Riley W, Stone A, et al. Initial item banks and first wave testing of the Patient-Reported Outcomes Measurement Information System (PROMIS) network: 2005-2008. *Journal of Clinical Epidemiology*. 2010;63:1179-1194.
- **160.** PROMIS. Adult Depression version 1.0 short form: a breif guide to the 8-item PROMIS Short Form v1.0-Depression 8b. 2012; <a href="http://assessmentcenter.net">http://assessmentcenter.net</a>.
- **161.** PROMIS. Adult satisfaction with participation in social roles profile short forms. 2013; Http://assessmentcenter.net.
- **162.** PROMIS. Adult physical function profile short forms. 2013; http://assessmentcenter.net.
- **163.** Cella D, Yount S, Rothrock N. The Patient-Reported Outcomes Measurement Information System (PROMIS): Progress of an NIH Roadmap Cooperative Group during its First Two Years. *Med Care*. 2007;45(5 Suppl):S3-S11.
- **164.** Sikorskii A, Given C, You M, Jeon S, Given B. Response analysis for multiple symptoms revealed differences between arms of a symptom management trial. *Journal of Clinical Epidemiology*. 2009;62(7):716-724.
- **165.** Given CW, Given BA, Sikorskii A, et al. Deconstruction of nurse-delivered patient self-management interventions for symptom management: factors related to delivery enactment and response. *Ann Behav Med.* Aug 2010;40(1):99-113.
- **166.** Jeon S, Given C, Sikorskii A, Given B. Do interference-based cut-points differentiate mild, moderate and severe levels of 16 cancer-related symptoms over time? *Journal of Pain and Symptom Management.* 2009;37(2):220-232.
- **167.** Bayliss EA, Ellis JL, Steiner JF. Seniors' self-reported multimorbidity captured biopsychosocial factors not incorporated into two other data-based morbidity measures. *Journal of Clinical Epidemiology*. 2009;62(5):550-557.
- **168.** Devilly GD, & Borkovec TD. Psychometric properties of the Credibility/Expectancy Questionnaire. *Journal of Behavior Therapy & Experimental Psychiatry*. 2000;31: 73-86.
- **169.** Wyatt GK. Complementary therapy utilization survey (unpublished instrument). East Lansing, MI: Michigan State University; 1993.
- **170.** Given C, Given B, Stommel M, Collins C, King S, Franklin S. The caregiver reaction assessment (CRA) for caregivers to persons with chronic physical and mental impairments. *Research in Nursing and Health.* 1992;15(4):271-283.
- **171.** PROMIS. Patient-Reported Outcomes Measurment Information System, Version 1.0 2010; <a href="https://www.nihpromis.org">www.nihpromis.org</a>. Accessed September 25, 2012.

- Wyatt G, Frambes D. Patient satisfaction with friend or family caregiver involvement. East Lansing, MI: College of Nursing, Michigan State University; 2012.
- **173.** Sikorskii A, Noble PC. Statistical Considerations in the Psychometric Validation of Outcome Measures. *Clin Orthop Relat Res.* May 4 2013.
- **174.** Kintner EK, Sikorskii A. Reliability and construct validity of the Participation in Life Activities Scale for children and adolescents with asthma: an instrument evaluation study. *Health Qual Life Outcomes*. 2008;6:43.
- **175.** Wyatt G, Sikorskii A, Wills CE. Development and Initial Validation of a Complementary and Alternative Medicine (CAM) Knowledge Instrument. *Journal of Nursing Measurement*. 2013;21(1):55-63.
- **176.** Sikorskii A, Melfi V, Gilliland D, Kaplan J, Ahn S. Quantitative literacy at Michigan State University: Development and initial evaluation of the assessment. *Numeracy.* 2011;4(2):Article 5.
- 177. Little R, Rubin M. Statistical Analysis with Missing Data. New York: Wiley and Sons; 1987.
- **178.** Hogan JW, Roy J, Korkontzelou C. Handling drop-out in longitudinal studies. *Statistics in Medicine*. 2004;23(9):1455-1497.
- 179. Shen C, Weissfeld L. Application of pattern-mixture models to outcomes that are potentially missing not at random using pseudo maximum likelihood estimation. *Biostatistics*. 2005;6(2):333-347.
- **180.** Given CW, Given BA. Symptom Management and Psychosocial Outcomes Following Cancer In: Oeffinger K, ed. *Submitted to Seminars in Oncology, Special Edition* 2013.
- **181.** Robbins JM. Optimal structured nested models for the optimal sequential decisions. In: Lin DY, Heagerty PJ, eds. *Proceedings of the Second Seattle Wymposium on Biostatistics*. New York, NY: Springer; 2004.
- **182.** Moodie EE, Richardson TS, Stephens DA. Demystifying optimal dynamic treatment regimes. *Biometrics.* Jun 2007;63(2):447-455.
- **183.** Murphy SA. A Generalization Error for Q-Learning. *J Mach Learn Res.* Jul 2005;6:1073-1097.
- **184.** Sutton RS, Barto AG. Reinforcement learning: An introduction. Cambridge, MA: MIT Press; 1998.
- **185.** Murphy SA. Optimal dynamic treatment regimes (with discussions). *Journal of the Royal Statistical Society, Series B.* 2003;65:331-366.
- **186.** Benjamini Y, Hochberg Y. Controlling the false discovery rate: A practical and powerful approach to multiple testing. *J of the Royal Statistical Society, Series B.* 1995;57(1):289-300.
- **187.** Benjamini Y, Yekutieli D. The control of the false discovery rate in multiple testing under dependency. *Annals of Statistics*. 2001;29(4):1165-1188.

**188.** Thissen D, Steinberg L, Kuang D. Quick and easy implementation of the Benjamini-Hochberg procedure for controlling the false positive rate in multiple comparisons. *Journal of Educational and Behavioral Statistics*. 2002;27(1):77-83.